CLINICAL TRIAL: NCT00608920
Title: SPECT Lymph Node Mapping to Define Nodal Clinical Target Volume in Patients With Prostate Cancer
Brief Title: Single Photon Emission Computed Tomography (SPECT) Lymph Node Mapping
Acronym: SPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-0772
Record Dates: First submitted 2008-01-02; First posted 2008-02-06 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: SPECT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPECT lymph node mapping (Experimental): 1. Diagnostic pelvic CT
  2. Nuclear tracer injection (Tc-99m) - same time as the ACCULOC seed implantation
  3. CT simulation (2 hours after prostate markers are placed)
  4. SPECT lymphoscintigraphy (first set of images 3-6 hours after injection and second set may be obtained 18-24 hours after injection)
  Interventions: Other: Single Photon Emission Computed Tomography (SPECT)

INTERVENTIONS:
Other: Single Photon Emission Computed Tomography (SPECT)

SUMMARY:
The purpose of this study is to determine if the planning of radiation treatment of prostate cancer patient can be made more precise by comparing currently planning techniques to an imaging technique called SPECT.

DETAILED DESCRIPTION:
Single photon emission computed tomography (SPECT) uses radioactive tracers and a scanner to record data that a computer constructs into two- or three-dimensional images. A small amount of a radioactive drug is injected into the body and a scanner is used to make detailed images of areas inside the body where the radioactive material is taken up by the cells. Using a gamma camera (a special kind of scanner), we can create a better picture of the lymph node region. We will compare these pictures to images from your CT scan, to help plan your therapy.

The research in this study involves seeing if it is feasible to use SPECT scanning procedures for the purpose of planning your radiation treatment. We hope that doing so will allow us to more accurately and precisely plan radiation treatment to potential sites of cancer, and avoid delivering too much radiation to normal

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven adenocarcinoma of the prostate
* Patients with at least one of the following high risk clinical features at the time of presentation:
* Extra-prostatic extension (on palpation or radiographic imaging)
* PSA ≥ 20
* Gleason Score ≥ 8
* Patients scheduled to receive prostatic and pelvic IMRT with ACCULOC® target localization
* Age > 18 years
* ECOG Performance Status ≤ 2
* Willing and able to sign informed consent document.-

Exclusion Criteria:

* History of radical prostatectomy
* History of prior pelvic radiation-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of using SPECT-LM | Completion of enrollment of all patients
  Safety: The study will be feasible if no more than 80% of patients experience the following complications: infection requiring hospitalization or IV antibiotics, urinary retention requiring placement of a Foley catheter, moderate or severe allergic reaction to Tc99.
  Efficacy: The study will be feasible if at least 80% of patients have at least one identifiable lymph node on SPECT-LM.

SECONDARY OUTCOMES:
Evaluate the extent to which current target delineation guidelines include actual lymphatic channels visualized on SPECT-LM in the study population. | Completion of enrollment of all patients
  1. Greatest radial distance of lymphatic channel volume from vessel wall contour
  2. Fraction of lymphatic channel volume, normal tissue volume, and critical structure volumes included in radial expansions from vessel wall

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Michalski, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu